CLINICAL TRIAL: NCT03819127
Title: Effects of Vildagliptin, a DPP-4 Inhibitor, in Elderly Diabetic Patients With Mild Cognitive Impairment
Brief Title: Vildagliptin in Older Adults With Diabetes and Mild Cognitive Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Enzo Saretto Dante Vicari, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/2015
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Vildagliptin; Tablets; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): metformin 1 g twice a day for 24 weeks
  Interventions: Drug: Metformin Pill
- Metformin plus vildagliptin (Experimental): metformin 1 g plus vildagliptin 50 mg twice a day for 24 weeks
  Interventions: Drug: Vildagliptin 50 MG Oral Tablet; Drug: Metformin Pill

INTERVENTIONS:
Drug: Vildagliptin 50 MG Oral Tablet
  Arms: Metformin plus vildagliptin
Drug: Metformin Pill

SUMMARY:
This study investigates the effect of vildagliptin, an inhibitor of the enzyme DPP-4, on the cognitive functioning of elderly diabetic patients with mild cognitive impairment (MCI) documented at mini mental state examination (MMSE).

In this prospective study, 60 diabetic elderly people were enrolled and divided according to their glycated hemoglobin (HbA1c) values in 2 groups: Group A, (HbA1c <7.5%, n=30) treated with metformin, and Group B (HbA1c >7.5%, n=30) treated with metformin plus vildagliptin. We evaluated MMSE, fasting plasma glucose (FPG) and HbA1c at baseline and after 24 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* age >65 years
* MMSE score ≥18 and ≤23
* diagnosis of diabetes mellitus

Exclusion Criteria:

* heart failure
* coronary heart disease
* stroke
* chronic kidney disease (G3 grade KDOQI)
* liver cirrhosis
* chronic respiratory failure
* depression evaluated by Geriatric Depression (GDS, GDS >15)
* diagnosis of dementia based on DSM 5 criteria
* anticholinesterase or memantine therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of cognitive decline | 24 weeks
  Mini Mental State Examination (MMSE) score from 0 (worse) to 30 points (better). Score ≥18 and ≤23 indicates mild cognitive impairment (MCI).

SECONDARY OUTCOMES:
Rate of Glycated hemoglobin (%) | 24 weeks
  Laboratory assessment of Glycated hemoglobin